CLINICAL TRIAL: NCT04915963
Title: Effect of a Single Mega-dose of Vitamin D3 Supplementation on Clinical Course in Non-deficient Patients Admitted in Intensive Care Unit
Brief Title: Vitamin D Supplementation in Intensive Care Unit Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Association Tunisienne d'Etude & de Recherche sur l'Athérosclérose (Other)
Collaborators: Faculty of Medicine of Tunis (Other); Rabta University Hospital (Unknown)
Responsible Party: Principal Investigator, Amani Kallel, Associate professor, Association Tunisienne d'Etude & de Recherche sur l'Athérosclérose
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HR-2015/08
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Dietary Supplements; Intensive Care Unit; Vitamin D Deficiency; Vitamin D Toxicity
Keywords: Critically ill; Intensive care unit; Vitamin D deficiencies
MeSH Terms: conditions — Vitamin D Deficiency; Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vitamin D group (Experimental): 170 patients receiving a single dose of 400,000 IU of VD3 (2 vials of 200,000 IU VD3; B.O.N., BOUCHARA RECORDATI) orally or through a nasogastric tube
  Interventions: Dietary Supplement: Vitamin D supplementation
- Placebo group (Sham Comparator): 170 patients receiving distilled water (2 vials of 1 ml distilled water) orally or through a nasogastric tube
  Interventions: Dietary Supplement: Vitamin D supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin D supplementation — Patients are randomized to receive vitamin D or placebo and followed up for 15 days at maximum to investigate the safety and clinical efficacy of the supplements

SUMMARY:
A randomized controlled trial is designed to investigate the safety and clinical efficacy of a mega dose of VD in patients admitted in intensive care unit (ICU). Patients will be randomly allocated to receive 400,000 IU of VD3 or placebo. They will be followed up until ICU discharge or death or the 15th day of ICU stay. Adverse events that occur during ICU stay is collected. Primary outcome is intensive care unit-acquired infection (ICU-AI), and secondary outcomes are septic shock, organ failure, and ICU-mortality. Plasma 25-hydroxyvitamin D is assessed at baseline and at the end of follow-up. Cox regression models will be applied to test how VD supplementation affects adverse outcomes while adjusting for confounders.

DETAILED DESCRIPTION:
The randomized controlled trial aimed to investigate the safety and clinical efficacy of a single mega dose of vitamin D (VD) in patients admitted at intensive care unit (ICU).

Study participants: VD deficient ICU patients

Criteria of inclusion, patients:

* newly admitted (within 24 hours)
* over eighteen,
* able to receive medication orally or through nasogastric tube
* expected to stay more than 72 hours in ICU.

Criteria for non-inclusion and exclusion, patients:

* lack of patient's or relatives' consent
* expected short life or ICU stay (<48 hours)
* sepsis at admission
* kidney, liver or intestinal disease
* hypercalcemia (total calcium>10.6 mg/dL)
* history of a disorder associated with hypercalcemia (cancer, tuberculosis, sarcoidosis, hyperparathyroidism, nephrolithiasis)
* treatment with immunotherapy or vitamin supplements within one year
* pregnant or breastfeeding women
* discharge from ICU or death within 72 hours of admission

Study protocol

Patients will undergo physical examination with calculation of acute physiology and chronic assessment II (APACHE II) and sequential organ failure assessment (SOFA) scores. They will be randomly assigned to either VD or placebo group after stratification on gender, age and APACHE II:

* VD group, 170 patients will receive a single dose of 400,000 IU of VD3 orally or through nasogastric tube
* Placebo group, 170 patients will receive distilled water orally or through nasogastric tube.

The patients will followed up until ICU discharge or death or the 15th day of ICU stay, whichever occurs first and adverse events that occurred during ICU stay were collected.

Primary outcome: intensive care unit-acquired infection (ICU-AI), defined as an infection of blood stream, lower respiratory tract, urinary tract, skin/soft tissue or gastrointestinal tract, which was not present within the first 48 hours of admission into the ICU.

Secondary outcomes: urinary calcium:creatinine ratio as surrogate for VD toxicity, septic shock, organ failure, ICU-mortality.

Plasma 25-hydroxyvitamin D (25-OHD) will be assessed at baseline and the end of follow-up using immunoassay.

Cox regression models will be applied to test how VD supplementation affects adverse events and ICU-mortality while adjusting for confounders.

Hypothesis. Recovering an adequate VD status might reduce poor outcome, especially infectious outcomes in ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* newly admitted (within 24 hours)
* over eighteen,
* able to receive medication orally or through nasogastric tube
* expected to stay more than 72 hours in ICU
* given consent

Exclusion Criteria:

* lack of patient's or relatives' consent
* expected short life or ICU stay (<48 hours)
* sepsis at admission
* kidney, liver or intestinal disease
* hypercalcemia (total calcium>10.6 mg/dL)
* history of a disorder associated with hypercalcemia (i.e., cancer, tuberculosis, sarcoidosis, hyperparathyroidism, nephrolithiasis)
* treatment with immunotherapy or vitamin supplements within one year
* pregnant or breastfeeding women
* discharge from ICU or death within 72 hours of admission

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Rate of intensive care unit-acquired infection (ICU-AI) | 15 days
  Infection of blood stream, lower respiratory tract, urinary tract, skin/soft tissue or gastrointestinal tract, which was not present within the first 48 hours of admission into the ICU, which occur during the ICU stay.

SECONDARY OUTCOMES:
urinary calcium:creatinine ratio | 15 days
  used as a surrogate for VD toxicity
Rate of septic shock | 15 days
  persisting hypotension requiring vasopressors to maintain a mean arterial pressure of<65 mm Hg and a serum lactate level >2 mmol/L despite adequate volume resuscitation .
Rate of organ failure | 15 days
  acute change in sequential organ failure assessment (SOFA) score of 2 points or greater secondary to infection
Rate of ICU-mortality | 15 days
  Death within the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Moncef Feki, Professor, Study Director — Rabta University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Thomas MK, Lloyd-Jones DM, Thadhani RI, Shaw AC, Deraska DJ, Kitch BT, Vamvakas EC, Dick IM, Prince RL, Finkelstein JS. Hypovitaminosis D in medical inpatients. N Engl J Med. 1998 Mar 19;338(12):777-83. doi: 10.1056/NEJM199803193381201. PMID 9504937
- [Background] Kvaran RB, Sigurdsson MI, Skarphedinsdottir SJ, Sigurdsson GH. Severe vitamin D deficiency is common in critically ill patients at a high northern latitude. Acta Anaesthesiol Scand. 2016 Oct;60(9):1289-96. doi: 10.1111/aas.12748. Epub 2016 Jun 12. PMID 27291260
- [Background] Leaf DE, Raed A, Donnino MW, Ginde AA, Waikar SS. Randomized controlled trial of calcitriol in severe sepsis. Am J Respir Crit Care Med. 2014 Sep 1;190(5):533-41. doi: 10.1164/rccm.201405-0988OC. PMID 25029202
- [Background] Amrein K, Schnedl C, Holl A, Riedl R, Christopher KB, Pachler C, Urbanic Purkart T, Waltensdorfer A, Munch A, Warnkross H, Stojakovic T, Bisping E, Toller W, Smolle KH, Berghold A, Pieber TR, Dobnig H. Effect of high-dose vitamin D3 on hospital length of stay in critically ill patients with vitamin D deficiency: the VITdAL-ICU randomized clinical trial. JAMA. 2014 Oct 15;312(15):1520-30. doi: 10.1001/jama.2014.13204. PMID 25268295
- [Background] Kempker JA, West KG, Kempker RR, Siwamogsatham O, Alvarez JA, Tangpricha V, Ziegler TR, Martin GS. Vitamin D status and the risk for hospital-acquired infections in critically ill adults: a prospective cohort study. PLoS One. 2015 Apr 7;10(4):e0122136. doi: 10.1371/journal.pone.0122136. eCollection 2015. PMID 25849649
- [Background] Ala-Kokko TI, Mutt SJ, Nisula S, Koskenkari J, Liisanantti J, Ohtonen P, Poukkanen M, Laurila JJ, Pettila V, Herzig KH; FINNAKI Study Group. Vitamin D deficiency at admission is not associated with 90-day mortality in patients with severe sepsis or septic shock: Observational FINNAKI cohort study. Ann Med. 2016;48(1-2):67-75. doi: 10.3109/07853890.2015.1134807. Epub 2016 Jan 22. PMID 26800186
- [Background] Quraishi SA, De Pascale G, Needleman JS, Nakazawa H, Kaneki M, Bajwa EK, Camargo CA Jr, Bhan I. Effect of Cholecalciferol Supplementation on Vitamin D Status and Cathelicidin Levels in Sepsis: A Randomized, Placebo-Controlled Trial. Crit Care Med. 2015 Sep;43(9):1928-37. doi: 10.1097/CCM.0000000000001148. PMID 26086941